# Statistical Analysis Plan (SAP)

CTN-0093: Validation of a Community Pharmacy-Based Prescription Drug Monitoring Program Risk Screening Tool

NCT039369

Document created July 17, 2019



# CTN-0093 Statistical Analysis Plan

# VALIDATION OF A COMMUNITY PHARMACY-BASED PRESCRIPTION DRUG MONITORING PROGRAM RISK SCREENING TOOL (PHARMSCREEN)

SAP Author: Ziji Yu, PhD

Senior Statistician: Ben Haaland, PhD

University of Utah Statistical Design and Biostatistics Center

June 17, 2019

## 1.0 STUDY DESIGN AND OBJECTIVES

## 1.1 STUDY DESIGN

This study is a one group, cross-sectional, validation study. Approximately 1,523 adults prescribed opioid medications will be recruited from one of 15 participating Kroger Pharmacies. Two sources of data will be obtained for this study. The first source is participants will complete self-report assessments via a secure on-line portal regarding contact; demographic; and behavioral and physical health information. The second source is the Narcotic Score (NS), referred to as the "NS metric" herein, which will be provided by Appriss Health.

# 1.2 STUDY OBJECTIVES

The goal of the study is to validate NS metric as Prescription Drug Monitoring Program-based instrument to discriminate between low, moderate, and high-risk opioid use disorder. The World Health Organization Alcohol, Smoking, and Substance Involvement Screening Test (WHO ASSIST) will be used as the gold standard instrument that defines patient risk levels. No intervention or hypothesis will be tested.

There are 2 statistical Aims in the project:

**Aim 1:** To assess the overall ability of NS metric to discriminate between opioid use risk levels and to determine cut-point thresholds for NS metric total score to classify patients into low, moderate, and high risk groups.

**Aim 2:** To validate the NS metric classifier (with selected cut-point threshold values from Aim 1 as a clinical measure to evaluate patients' opioid risk level, with WHO ASSIST as the gold standard to which the NS metric is compared.

Other exploratory statistical Aims include:

- To explore the association between NS metric and other indicators of opioid use risk, such as: the Tobacco, Alcohol, Prescription medication and other Substances (TAPS) Tool; a positive misuse indication from the Prescription Opioid Misuse Index (POMI); and history of opioid overdose.
- To collect validity data on the TAPS tool in a large sample of individuals filling opioid pain medications.

#### 2.0 GENERAL DEFINITIONS

## 2.1 DEFINITION OF STUDY POPULATION

# 2.1.1 ALL ENROLLED SUBJECTS POPULATION

The enrolled subjects population (ENR) will contain all participants who provide informed consent for this study and are deemed as meeting the inclusion/exclusion criteria. ENR will be used to summarize subject disposition.

## 2.1.2 COMPLETER POPULATION

A participant is considered as a completer if all of the participant's electronic Case Report Forms (eCRFs) have been completed, although it is possible that some questions on the eCRFs may not be answered. The completer population will be used as the main analysis population.

# 2.2 DEFINITION OF ASSESSMENTS

## **2.2.1 NS METRIC**

Appriss Health has developed the NS metric, which uses PDMP data on prescription opioid and benzodiazepine use and aberrant drug behavior (e.g., multiple providers, pharmacies) to compute a score quantifying the extent of the patient's risk in relation to all prescription opioid users. The NS metric is a continuous indicator on a 000-999 scale, with the last digit representing active number of opioid prescriptions (those with ≥9 prescriptions coded as 9) and the first two numbers representing a composite risk score. Higher scores indicate increased risk for adverse opioid-related outcomes (e.g., overdose). See CTN-0093 Protocol Study Assessments section for details on score composition.

# 2.2.2 WHO ASSIST

The WHO ASSIST opioid use risk domain will be used as the gold standard to which the NS metric will be compared. The WHO ASSIST opioids domain is a continuous indicator on a 0-20 scale, with the 0-0.5 range representing low risk, the 0.5-14.5 range representing moderate risk, and the 14.5-20 range representing high risk. <sup>1</sup> The WHO ASSIST has demonstrated criterion, construct, concurrent, and discriminant validity. <sup>1</sup>

### **2.2.3 TAPS**

The TAPS Tool consists of a 5-item screening for tobacco use, unhealthy alcohol use, prescription medication misuse, and illicit substance use. Positive reports on the screener result in respondents subsequently being asked 9 additional substance specific items. Scoring on the TAPS Tool involves summing respondents' answers to the substance specific questions, resulting in a 0-3 ordinal score for each drug (0=No use in the past 3 months; 1= problem use; 2= higher risk). The TAPS Tool has demonstrated concurrent validity. <sup>2</sup> This measure will be captured in order to provide additional information regarding its psychometric properties compared to the WHO ASSIST.

## 2.2.4 OTHER MEASUREMENTS

Covariates known to be correlated with opioid use severity will also be captured. These covariate measures will include: opioid medication misuse, pain severity, general health status, depression, overdose frequency history.

A list of study measurements and domains of interest are summarized in **Table 1**:

| Table 1. Study | Measures | | |
|---|---|---|---|
| | | No. of | Min. to |
| Domain | Name | Items | Complete |
| Opioid use | WHO Alcohol, Smoking and | 8 | <b>≤</b> 5 |
| severity | Substance Involvement Screening Test | | |
| | (ASSIST): Opioid Items <sup>1</sup> | | |
| | WHO Alcohol, Smoking and | 16 | <b>≤</b> 5 |
| | Substance Involvement Screening Test | | |
| | (ASSIST): Adapted heroin and prescription opioid | | |
| | items <sup>3*</sup> | | |
| | Tobacco, Alcohol, Prescription Medication, and Other | 2-4 | ≤1 |
| | Substance Use (TAPS) 1 / 2 Tool: Prescription drug | | |
| | and prescription opioid items <sup>2</sup> | | |
| | Tobacco, Alcohol, Prescription Medication, and Other | 2-4 | ≤1 |
| | Substance Use (TAPS) 1 / 2 Tool: <i>Illicit drug and</i> | | |
| | heroin items <sup>2</sup> | | |
| Opioid | Prescription Opioid Misuse Index <sup>4</sup> | 6 | <b>≤</b> 5 |
| medication | | | |
| misuse | | | |
| Opioid | Overdose Experiences, Self and Witnessed—Drug | 1 | ≤1 |
| overdose | (OESWD) <sup>5</sup> | | |
| Non-opioid | WHO Alcohol, Smoking and | 8-72 | 5-15 |
| drug use | Substance Involvement Screening Test | | |
| severity | (ASSIST): Non-opioid drug use items <sup>1</sup> | | |
| | Tobacco, Alcohol, Prescription Medication, and Other | 12-25 | <b>≤</b> 5 |
| | Substance Use (TAPS) 1 / 2 Tool: Non-opioid items <sup>2</sup> | | |
| Depression | Patient Health Questionnaire-2 <sup>6</sup> | 2 | ≤1 |
| Physical | Short Form-12: General health subscale <sup>7</sup> | 1 | ≤1 |
| Health | Brief Pain Inventory <sup>8</sup> | 8 | ≤5 |
| Demographics | PhenX demographics: age, education, gender, race, | 10 | <5 |
| | ethnicity, health insurance, employment, marital status | | |
| | Totals: | 76-157 | 40-50 |

<sup>\*</sup> The adapted heroin and prescription opioid items will not be employed in the a priori analyses.

# 3.0 STATISTICAL CONSIDERATION

# 3.1 MULTICENTER STUDIES

This study will be conducted by multiple investigators at multiple Universities; however, these data will be captured in a single REDCap data system. Descriptive statistics on demographic, other characteristics, and clinical measurements of interests (described in Section 2.2) will be presented by pharmacy recruitment site and between site differences will be examined.

# 3.2 DATA MANAGEMENT

Throughout the data collection phase of the study, the OVN and University of Utah teams will

collaborate to share a cleaned identified datasets with Appriss Health. Using the patient name, contact information, survey timestamp, and store location; Appriss will deterministically match NS metric data with the final dataset and share a merged dataset with OVN and the University of Utah for analyses. It is important to note that given the privacy of the survey response method (i.e., self-report outside of the pharmacy setting), we anticipate participant responses will have less measurement error (e.g., less social desirability bias). Thus, we anticipate our participant responses will more accurately relate to objective PDMP information than interviewer administered or pharmacy-based surveys.

# 3.3 DISPOSITION

The number and percentages of screened and enrolled subjects as well as subjects who complete all eCRFs will be presented based on ENR.

## 3.4 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISITCS

Demographic data and other baseline characteristics will be summarized using descriptive statistics for the Completers Population and ENR. Demographic and other baseline characteristics include, but are not limited to:

- Age (years) calculated relative to date of submitted e-consent
- Education
- Birth gender
- Race
- Ethnicity
- Health Insurance
- Employment
- Marital status

# 3.5 STATISTICAL METHODS

The Completer Population will be randomly split into training data set and testing data set with a 1:1 ratio, stratified by WHO ASSIST risk levels. The training data set will be used to select cutpoints for NS metric risk levels, and testing data set will be used to address statistical Aim 2, validating the selected cut-points. The proposed approach allows us to assess the predictive ability of the NS metric classifier with an independent testing data set and avoid potentially overfitting. All analyses will be performed both overall and within sex specific subpopulations, to examine sex difference in discrimination, selected cut-points, and agreement between measures.

Summary statistics will be provided for the following clinical assessments for the population, by gender subpopulation, by pharmacy recruitment sites.

- NS Metric
- WHO ASSIST
- TAPS
- OESWD
- Prescription Opioid Misuse Index
- PHQ-2
- SF-12
- Brief Pain Inventory

Statistical Aim 1 - To assess the ability of NS metric to discriminate between opioid use risk groups and to determine cut-off points for NS metric total score.

To assess the ability of NS metric to discriminate between opioid use risk groups:

The discriminative validity of an instrument concerns its ability to discriminate between known groups. In the project, the known groups are the low risk, moderate risk, and high risk groups as defined by WHO ASSIST opioid domain (0-0.5 range=low risk, 0.5-14.5 range=moderate risk, and 14.5-20 range=high risk).

A receiver operating characteristics (ROC) analysis<sup>10</sup> will be conducted to 1) assess the overall discriminative ability of NS metric score as a clinical risk assessment instrument, 2) select cutpoint threshold values to define low, moderate, and high risk groups with NS metric.

Area under the ROC curve (AUC) values will be used to determine the overall discriminating ability of NS metric. AUC is an overall performance measurement for the classification of an instrument at various threshold settings, and it tells how much the classifier is capable of distinguish between classes. The following scale will be used for the evaluation: <0.70=poor,  $\ge 0.70=$ fair,  $\ge 0.80$  good  $\ge 0.9=$ excellent.

The study will be powered to the least prevalent but most severe condition among potential patients. Based on the allocation ratio of the national rate of prescription opioid use disorder (POUD) among those prescribed opioid medications in the last year, the prevalence of POUD is 2.1%. A sample of approximately 1,523 (32 positive group) achieves 97.68% power to detect a difference of 0.2 between the area under the ROC curve (AUC) under the null hypothesis of 0.5 and the alternative hypothesis of 0.7 using a two-sided z-test at a significance level of 0.050.

The Completer Population (both training and testing set) will be used to assess the overall discrimination ability of NS metric.

*To determine cut-point threshold values for NS total score:* 

The objective is to select the optimal cut-points threshold for NS metric to define low, moderate and high risk groups. We will use a hybrid framework where we can make use of the data driven methods to support the clinician's final decision making. Only the training data set will be used in this portion of analysis.

In the first step, the solution space (a subset of optimum choices of cut-point threshold values) will be identified with the following grid search approach: for each pair of risk groups, for example, low risk vs moderate risk, calculate the following performance measurements for each possible cut-point threshold value:

• Sensitivity (SE)

$$SE = \frac{True \ Positive \ Rate}{True \ Positive \ Rate + False \ Negative \ Rate}$$

• Specificity (SP)

$$SP = \frac{True \text{ Negative Rate}}{True \text{ Negative Rate} + False \text{ Postive Rate}}$$

- Positive Predictive Value (PPV): probability that the risk level is present (based on WHO ASSIST) when the result with NS metric is positive.
- Negative Predictive Value (NPV): probability that the risk level is not present (based on WHO ASSIST) when the test result with NS metric is negative.
- Youden's index:

Youden's Index = 
$$SE + SP - 1$$

Youden's index, a metric that summarizes both false positive and false negative misclassification rates with equal weights, will be used as primary evaluation criteria to compare classification performance across scenarios with different cut-points threshold values. A solution space, i.e. a set of cut-point threshold values with highest Youden's Index, will be selected. For example, the selected solution space of low risk vs moderate risk cut-point threshold is 10-30, which gives the highest 10% Youden's Index among all possible choices (0-999). See **Table 2** as an example of grid search result:

| Table 2: Grid sear | ch result for tl | reshold | value of m | oderate v | s high ris | ks | |
|---|---|---|---|---|---|---|---|
| Possible | Youden's | SE | SP | PPV | NPV | Rank of | Flag for |
| Threshold values | Index | | | | | Youden's | solution space |
| for high risk vs | | | | | | Index | |
| moderate risk | | | | | | | |
| 0 | XXX | XXX | XXX | XXX | XXX | | |
| ••• | | | | | | | |
| 511 | XXX | XXX | XXX | XXX | XXX | 10/1000 | Yes |
| 512 | XXX | XXX | XXX | XXX | XXX | 100/1000 | Yes |
| 513 | XXX | XXX | XXX | XXX | XXX | 200/1000 | No |
| ••• | | | | | | | |
| 999 | XXX | XXX | XXX | XXX | XXX | | |

In the second step, the final optimal cut-points threshold values will be selected from the solution space, with clinical justification such that the balance between sensitivity and specificity is achieved. For example, a cut-off point of 20 is selected for low risk vs moderate risk group based upon clinician's justification. This framework will integrate clinical knowledge into purely data-driven techniques.

Assuming the acceptable SE and SP are 0.8 for both cutoffs (low vs moderate/high and low/moderate vs high), with a sample size of 750 patients in the training data set, the width of 95% confidence intervals of SE and SP estimations are 0.026 and 0.056 for the classification cutoffs that predict low risk vs moderate/high (prevalence 82.9% vs 17.1%). For predicting low/moderate risk vs high risk (prevalence 2.1% vs 97.9%), the width of confidence intervals for SE and SP are 0.143 and 0.024, respectively. The narrow confidence intervals imply relatively high precision for the SE and SP estimations, which will be used to support clinicians' decision making.

The final selected cut-points threshold values will be validated with an independent testing data set in Aim 2.

Statistical Aim 2 – To validate discriminative ability of NS metric (with the established risk levels of low, moderate, and high) as a clinical measure to evaluate opioid use risk level.

The second primary aim of the project is to evaluate the concurrent validity of the NS metric with the established risk levels of low, moderate, and high. Classification accuracy will be evaluated with an independent testing data set, and WHO ASSIST will be used as the gold standard to define actual risk levels for patients. The agreement level of risk groups defined by NS metric and WHO ASSIST will be descriptively summarized with a confusion matrix, see **Table 3**. Each row of the matrix represents the instances and percentages in a predicted risk level while each column represents the instances in an actual risk level.

| Table 3. Co | nfusion matrix | | | |
|---|---|---|---|---|
| | | Actual risk levels defined by WHO ASSIST | | |
| | | Low | Moderate | High |
| Predicted | | risk level | risk level | risk level |
| risk levels | Low risk level | XXX(XX.XX%) | XX(XX.XX%) | XX(XX.XX%) |
| defined by | Moderate risk level | XX(XX.XX%) | XX(XX.XX%) | XX(XX.XX%) |
| NS metric | High risk level | XX(XX.XX%) | XX(XX.XX%) | XX(XX.XX%) |

Cohen's Kappa Coefficient<sup>11,12</sup> will be used to evaluate agreement between the two metrics. The following scale will be used to assess level of agreement: 0-0.2=slight, 0.21-0.4=fair, 0.41-0.6=moderate, 0.61-0.8=substantial, and 0.81-1=near perfect. We expect the NS metric will demonstrate at least moderate (≥0.40) agreement with the gold-standard risk categories, and a sample size of 750 patients and prevalence of 2.1% (for high risk level) will achieve 99.8% power with a significance level of 0.05 in a test of H0: Kappa ≤ 0.4 vs. H1: Kappa > 0.4. Agreement between NS metric and WHO ASSIST will also be evaluated via Spearman Correlation<sup>13</sup> based upon risk levels (1 for low risk, 2 for moderate risk, and 3 for high risk for both NS metric and WHO ASSIST). The following scale will be used to assess level of agreement: 0-0.3 = low degree, 0.3-0.5 = moderate degree, 0.5-1 = high degree.

An ordinal logistic regression model<sup>14</sup> will be built to estimate the magnitude of association between the metrics, while controlling for other relevant risk factors. In the ordinal logistic regression, WHO ASSIST risk levels will be considered as response variable, and regression covariates will include NS metric, and other relevant indicators known to be associated with opioid-related risk, including: sex, pain, general health status, depression, and substance use history (**Table 1**). The association between WHO ASSIST and NS metric will be estimated by odds ratios, and Wald statistics will be used to examine the association at a 0.05 significance level.

# Exploratory Statistical Aim 1: To validate TAPS tool using WHO ASSIST as gold standard.

The TAPS tool is rapidly becoming recognized as a high quality substance use screener for outpatient health care settings. Given the somewhat limited opioid using sample in the main outcomes study (≤5% for prescription opioids; <4% for heroin\*), the current study offers an important opportunity to further validate this instrument in a novel outpatient setting, community pharmacy, among a large opioid using population.

The performance of TAPS Tool will be evaluated relative to WHO ASSIST. We plan to compare subjects' responses to each substance of TAPS Tool with their responses to the corresponding domains of WHO ASSIST. The TAPS tool has four domains, and WHO ASSIST has 9 domains. Domains on the ASSIST will be combined with those of the TAPS Tool, see Table 4 for details:

Table 4: combinations of substances for WHO ASSIST

| | | | TAPS 1 | (past 12 mont | ths) |
|---|---|---|---|---|---|
| | | Tobacco | Alcohol | Illicit Drug | Prescribed<br>Medication |
| | Tobacco products (cigarettes, chewing tobacco, cigars, etc.) | Х | | | |
| | Alcoholic beverages (beer, wine, liquor, etc.) | | Х | | |
| | Cannabis (marijuana, pot, weed, hash, etc.) | | | X | |
| (s) | Cocaine (coke, crack, etc.) | | | X | |
| 3 month | Amphetamine type stimulants (speed, diet pills, ecstasy, methamphetamine, crystalmeth, etc.) | | | Х | Х |
| oast | Inhalants (nitrous, glue, poppers, etc.) | | | Х | |
| ASSIST (past 3 months) | Sedatives or sleeping pills (Valium,<br>Rohypnol, Ativan, Xanax, Klonopin, GHB,<br>etc.) | | | | Х |
| • | Hallucinogens (LSD, acid, mushrooms, PCP, Special K, etc.) | | | Х | |
| | Opioids (heroin, morphine, methadone, codeine, buprenorphine, suboxone, Oxycontin, Percocet, Vicodin, etc. | | | Х | Х |
| | Other (K2, Spice, Synthetic spice, Synthetic marijuana) | | | Х | |

The level of agreement between TAPS tool with the established risk levels of low, moderate and high on the WHO ASSIST will be evaluated with similar methods as described in Aim 2: ROC analysis will be used to examine concordance between each domain of the TAPS Tool and the corresponding clustered domain of WHO ASSIST. Risk levels of the WHO ASSIST for each clustered domain are defined as follow:

- WHO ASSIST Tobacco Domain:
  - Moderate and High risk >3
  - Low risk  $\leq$  3
- WHO ASSIST Alcohol Domain:
  - o Moderate and High risk >10
  - Low risk  $\leq 10$

- WHO ASSIST Illicit Drug Domain:
  - Moderate and High risk >3
  - Low risk  $\leq$  3
- WHO ASSIST Prescribed Medication Domain:
  - Moderate and High risk >3
  - Low risk  $\leq 3$ .

For each of these binary risk categories, Area under the ROC curve (AUC) values will be used to determine the overall discriminating ability of TAPS tool on each of the 4 domains.

Table) and the following statistical measurements of agreement, all with their respective 95% confidence intervals will be provided: Spearman correlation coefficient, Goodman and Kruskal's Gamma, and Kendall rank correlation coefficient. A logistic regression model will be built to estimate the magnitude of association between the metrics, while controlling for other relevant risk factors.

| Table 5. C | Table 5. Confusion matrix for Alcohol Domain | | | | | |
|---|---|---|---|---|---|---|
| | | | TAPS Tool observation | | | |
| | | 0 | 1 | 2 | 3 | 4 |
| Predicted | Low risk level | XX | XX | XX | XX | XX |
| risk | | (XX.XX%) | (XX.XX%) | (XX.XX%) | (XX.XX%) | (XX.XX%) |
| levels | | , , | | , , | · | , |
| defined | High/ | XX | XX | XX | XX | XX |
| by WHO | moderate risk | (XX.XX%) | (XX.XX%) | (XX.XX%) | (XX.XX%) | (XX.XX%) |
| ASSIST | level | | | | | |

Exploratory Statistical Aim 2: To assess the association between the NS metric and other measurements of opioid misuse.

In this exploratory aim, we will assess the relationship between the NS metric with the established risk levels of low, moderate and high risk and 1) ordinal prescription and heroin use scores from the TAPS Tool (prescribed medication and heroin domains), 2) a positive misuse indication from (POMI), and 3) overdose frequency history.

Risk levels will be defined as follow:

- TAPS Tool prescribed medication domain:
  - o High risk≥2;
  - o Low risk<2.

- POMI:
  - High risk  $\geq 2$ ;
  - Low risk <2.
- Overdose Frequency History OESWD domain:
  - Any Overdose >0;
  - $\circ$  No Overdose = 0.

We will likewise employ the above described statistical analyses for Exploratory Aim 1 and assess the association and agreement level between NS metric and the TAPS Tool, POMI, and Overdose Frequency History with the:

- Confusion table;
- AUC of ROC analysis;
- Spearman Correlation Coefficient;
- Goodman and Kruskal's Gamma;
- Kendall rank correlation coefficient;
- Ordinal Logit Regression.

# **Exploratory Statistical Aim 3: To validate definition of NS metric.**

In this section, we will validate the definition of NS metric and test if the third digit of NS metric (number of opioid prescription) is informative. We will examine an alternative definition of NS metric, named as NS metric v2, which consists of only the first two numbers of original NS metric, which ranges 00-99. Descriptive analyses will be conducted and correlation between NS metric and NS metric v2 will be examined with Spearman Correlation Coefficients. We will repeat the planned training/validation analyses in the primary analysis and compare the discriminative ability of NS metric v2 vs. NS metric. We expect the predictive power of NS metric v2 is lower than that of NS metric, which implies the 3rd digit in NS metric original definition is predictive. We will also repeat the training/validation analysis within each subgroup of patients with same numbers of opioid prescriptions. The overall discriminate ability for NS metric 2, described by average misclassification rate across subgroups, will be compared with primary analyses results. It is expected that the prediction accuracy is comparable, which implies the "opioid prescription number" information is well represented by the third digit of original NS metric definition.

# 3.6 EXAMINATION OF SUBGROUPS

Subgroup analyses will be conducted on the primary and exploratory aims for the following groups:

• Gender: male and female.

For the subgroup analyses, all completers in each subpopulation will be randomly split into training data set and testing data set with a 1:1 ratio, stratified by WHO ASSIST risk levels. The cut-off threshold values will be selected using similar methods as described in Aim 1 for each subgroup and validated using similar methods as described in Aim 2, with the testing set for the corresponding subgroup. We will compare the selected threshold values and their discriminative ability between subgroups, see **Table 6** for details. *It should be noted* that the study is *not* designed to detect certain agreement level between metrics with high statistical power within any subgroup.

| | nary table that compares disc<br>t-off threshold between 2 gen | | | |
|---|---|---|---|---|
| go.u.s | | Female | Male | Overall |
| AUC of ROC | Low risk vs Moderate risk | | | |
| | Moderate risk vs high risk | | | |
| NS Metric | Low risk vs Moderate risk | | | |
| cut-off values | Moderate risk vs high risk | | | |
| | Validation of select | ed cut-off val | ues | |
| Kappa coefficient | | | | |
| Spearman Correlation Coefficient | | | | |
| Goodman and Kruskal's Gamma | | | | |
| Kendall rank correlation coefficient | | | | |
| Odds ratio from | ordinal logit regression | | | |

# 3.7 MISSING DATA

The completer population, defined as participants who complete all opioid outcome score contributing items on the WHO ASSIST and TAPS tool, will be used for the main analysis. Completers also must have a NS metric score. As a result of the one-time cross-sectional nature of this study, participant attrition is not a concern. Rubin's multiple imputation approach will be used to impute missing covariates but missing outcome data will not be imputed.<sup>15</sup>

# 3.8 OUTPUT PRESENTATION

APPENDIX 1 shows conventions for presentation of data in outputs. The tables, figures, and listings (TFL) shells provided with this SAP describe the presentations for this study and therefore the format and content of the summary tables, figures and listings to be provided by SDBC Statisticians.

# 3.9 SOFTWARE

All analyses performed by the SDBC will use R 3.4.4 for windows software.

# APPENDIX 1 TABLES, FIGURE AND LISTING SHELLS

| Proposed Tables, Figur | res and Listings | | |
|---|---|---|---|
| Section | Table/Figure | Analysis | Title |
| | # | Population | |
| Enrollment and | Table 1.1 | ENR | Summary of Subject Disposition |
| Participant Status | Table 1.2 | ENR | Summary of Subject Disposition by Gender |
| | Table 1.3 | СР | Summary of Training/Testing Random Split, |
| | | | Overall and by Gender |
| Baseline | Table 2.1 | CP | Summary of Baseline Demographics |
| Demographics | Table 2.2 | CP | Summary of Baseline Demographics by Gender |
| | Table 2.3 | CP | Summary of Baseline Demographics by |
| | | | Investigation Site |
| Summary of Clinical | Table 3.1 | CP | Descriptive summary of WHO ASSIST |
| Assessment | Table 3.2 | CP | Descriptive summary of WHO ASSIST, by |
| | | | Gender |
| | Table 3.3 | CP | Descriptive summary of WHO ASSIST, by |
| | | | Investigation site |
| | Table 3.4 | CP | Descriptive summary of NS Metric |
| | Table 3.5 | CP | Descriptive summary of NS Metric, by Gender |
| | Table 3.6 | CP | Descriptive summary of NS Metric, by |
| | | | Investigation site |
| | Table 3.7 | CP | Descriptive summary of TAPS Tool |
| | Table 3.8 | CP | Descriptive summary of TAPS Tool, by Gender |
| | Table 3.9 | CP | Descriptive summary of TAPS Tool, by |
| | | | Investigation site |
| | Table 3.10 | CP | Descriptive summary of POMI Tool |
| | Table 3.11 | CP | Descriptive summary of POMI Tool, by Gender |
| | Table 3.12 | CP | Descriptive summary of POMI Tool, by |
| | | | Investigation site |
| | Table 3.13 | CP | Descriptive summary of OESWD |
| | Table 3.14 | CP | Descriptive summary of OESWD, by Gender |
| | Table 3.15 | CP | Descriptive summary of OESWD, by |
| | T 11 2 16 | C.D. | Investigation site |
| | Table 3.16 | CP | Descriptive summary of Prescription Opioid |
| | T 11 2 17 | CD | Misuse Index |
| | Table 3.17 | CP | Descriptive summary of Prescription Opioid |
| | Tol-1- 2 10 | CD | Misuse Index, by Gender |
| | Table 3.18 | CP | Descriptive summary of Prescription Opioid Migues Index, by Investigation site |
| | Table 3.19 | СР | Misuse Index, by Investigation site |
| | | | Descriptive summary of PHQ-2 |
| | Table 3.20 | CP CP | Descriptive summary of PHQ-2, by Gender |
| | Table 3.21 | CP | Descriptive summary of PHQ-2, by Investigation site |
| | Table 3.22 | CD | |
| | 1 able 3.22 | CP | Descriptive summary of SF12 |

| Section | Table/Figure | Analysis<br>Population | Title |
|---|---|---|---|
| | Table 3.23 | CP CP | Descriptive summary of SF12, by Gender |
| | Table 3.24 | CP | Descriptive summary of SF12, by Investigation |
| | 1 4010 5.21 | CI | site |
| | Table 3.25 | CP | Descriptive summary of Brief Pain Inventory |
| | Table 3.26 | CP | Descriptive summary of Brief Pain Inventory, by |
| | 1 5 . 2 . 5 | | Gender |
| | Table 3.27 | СР | Descriptive summary of Brief Pain Inventory, by |
| | | | Investigation site |
| Results for Aim 1 | Figure 3.1 | CP | NS metric ROC curve for discriminating high risk |
| | | | vs moderate risk opioid misuse patients defined |
| | | | by WHO ASSIST opioid items. |
| | Figure 3.2 | CP | NS metric ROC curve for discriminating |
| | | | moderate risk vs low risk opioid misuse patients |
| | | | defined by WHO ASSIST opioid items. |
| | Figure 3.3 | CP | NS metric ROC curve for discriminating high risk |
| | | | vs moderate risk opioid misuse patients defined |
| | | | by WHO ASSIST opioid items, by gender |
| | Figure 3.4 | CP | NS metric ROC curve for discriminating |
| | | | moderate risk vs low risk opioid misuse patients |
| | | | defined by WHO ASSIST opioid items, by |
| | TD 11 0.5 | CP | gender |
| | Table 3.5 | CP | Summary of AUC of ROC curve |
| | Table 3.6 | CP | Summary of AUC of ROC curve, by gender |
| | Table 3.7 | CP - | Summary of grid search: ROC analysis results for |
| | | Training | all possible cut-off threshold values of high risk |
| | Table 3.8 | CP - | vs moderate risk with NS metric. |
| | 1 able 5.8 | | Summary of grid search: ROC analysis results for |
| | | Training | all possible cut-off threshold values of moderate risk vs low risk with NS metric. |
| | Table 3.9 | CP - | Summary of grid search: ROC analysis results for |
| | 1 aoic 3.7 | Training | all possible cut-off threshold values of high risk |
| | | Training | vs moderate risk with NS metric by gender |
| | Table 3.10 | CP - | Summary of grid search: ROC analysis results for |
| | 14616 5110 | Training | all possible cut-off threshold values of moderate |
| | | 8 | risk vs low risk with NS metric by gender |
| | Figure 3.11 | CP - | NS metric ROC curve for discriminating high risk |
| | | Training | vs moderate risk opioid misuse patients defined |
| | | C | by WHO ASSIST opioid items, with training data |
| | | | set. |
| | Figure 3.12 | CP - | NS metric ROC curve for discriminating |
| | | Training | moderate risk vs low risk opioid misuse patients |
| | | | defined by WHO ASSIST opioid items, with |
| | | | training data set. |
| | Figure 3.13 | CP - | NS metric ROC curve for discriminating high risk |

| Section | Table/Figure # | Analysis<br>Population | Title |
|---|---|---|---|
| | | Training | vs moderate risk opioid misuse patients defined<br>by WHO ASSIST opioid items, with training data<br>set, by gender. |
| | Figure 3.14 | CP -<br>Training | NS metric ROC curve for discriminating moderate risk vs low risk opioid misuse patients defined by WHO ASSIST opioid items, with training data set, by gender. |
| | Figure 3.15 | CP-<br>Training | Plot of Kappa Coefficient for NS metric vs WHO<br>Assist, for all possible threshold values in<br>selected solution space |
| | Figure 3.16 | CP -<br>Training | Plot of Kappa Coefficient for NS metric vs WHO Assist, for all possible threshold values in selected solution space, by gender |
| | Figure 3.17 | CP -<br>Training | Plot of Spearman Correlation Coefficient for NS metric vs WHO Assist, for all possible threshold values in selected solution space |
| | Figure 3.18 | CP -<br>Training | Plot of Spearman Correlation Coefficient NS metric vs WHO Assist, for all possible threshold values in selected solution space, by gender |
| | Figure 3.19 | CP -<br>Training | Plot of Specificity and Sensitivity, for all possible high vs moderate risk threshold in solution space |
| | Figure 3.20 | CP-<br>Training | Plot of Specificity and Sensitivity, for all possible moderate risk vs low risk threshold in solution space |
| | Figure 3.21 | CP -<br>Training | Plot of Specificity and Sensitivity, for all possible high vs moderate risk threshold in solution space, by gender |
| | Figure 3.22 | CP-<br>Training | Plot of Specificity and Sensitivity, for all possible moderate risk vs low risk threshold in solution space, by gender |
| | Figure 3.23 | CP -<br>Training | Plot of Positive Predictive Value and Negative<br>Predictive Value, for all possible high vs<br>moderate risk threshold in solution space |
| | Figure 3.24 | CP-<br>Training | Plot of Positive Predictive Value and Negative<br>Predictive Value, for all possible moderate vs<br>mild risk threshold in solution space |
| | Figure 3.25 | CP-<br>Training | Plot of Positive Predictive Value and Negative<br>Predictive Value, for all possible high vs<br>moderate risk threshold in solution space, by<br>gender |
| | Figure 3.26 | CP -<br>Training | Plot of Positive Predictive Value and Negative<br>Predictive Value, for all possible moderate vs<br>mild risk threshold in solution space, by gender |
| | Table 3.27 | CP - | Summary of ROC analysis result and Correlation |

| Section | Table/Figure | Analysis<br>Population | Title |
|---|---|---|---|
| | # | Training | Analysis result for the selected cut-off threshold value of NS metric, high vs moderate risk classification and moderate vs low risk classification |
| Results for Aim 2 | Table 4.1 | CP -<br>Testing | Confusion Table for NS metric with established cut-off threshold vs WHO ASSIST |
| | Table 4.2 | CP -<br>Testing | Confusion Table for NS metric with established cut-off threshold vs WHO ASSIST, by gender |
| | Table 4.3 | CP -<br>Testing | Summary of Kappa Coefficient and Correlation<br>Analysis Results, WHO ASSIST vs NS metric<br>(with established cut-off value from Aim 1) |
| | Table 4.4 | CP -<br>Testing | Summary of Kappa Coefficient and Correlation<br>Analysis Results, WHO ASSIST vs NS metric,<br>by gender (with established cut-off value from<br>Aim 1) |
| | Table 4.5 | CP -<br>Testing | Summary of ordinal logit regression results (with established cut-off value from Aim 1) |
| | Table 4.8 | CP -<br>Testing | Summary of ordinal logit regression results, by gender (with established cut-off value from Aim 1) |
| Results for<br>Exploratory Aim 1 | Table 5.1 | СР | TAPS Tool ROC curve for discriminating high risk vs low risk groups defined by WHO ASSIST, by domains (Tobacco, Alcohol, Illicit Drug, Prescribed Medication) |
| | Table 5.2 | СР | TAPS Tool ROC curve for discriminating high risk vs low risk groups defined by WHO ASSIST, by domains (Tobacco, Alcohol, Illicit Drug, Prescribed Medication), by gender |
| | Table 5.3 | CP | Summary of AUC of ROC curve for each domain |
| | Table 5.4 | CP | Summary of AUC of ROC curve for each domain by gender |
| | Table 5.5 | СР | Confusion Table for TAP Tool vs WHO ASSIST, for each domain |
| | Table 5.6 | CP | Confusion Table for TAP Tool vs WHO ASSIST, for each domain, by gender |
| | Table 5.7 | CP | Summary of Kappa Coefficient and Correlation<br>Analysis Results, WHO ASSIST vs TAP Tools<br>for each domain |
| | Table 5.8 | CP | Summary of Kappa Coefficient and Correlation<br>Analysis Results, WHO ASSIST vs TAP Tools<br>for each domain, by gender |
| | Table 5.9 | СР | Summary of ordinal logit regression results for each domain |
| | Table 5.10 | CP | Summary of ordinal logit regression results for |

| Section | Table/Figure | Analysis<br>Population | Title |
|---|---|---|---|
| | π | 1 opulation | each domain, by gender |
| Results for Exploratory Aim 2 – explore association | Table 6.1.1 | CP | Confusion Table for NS metric with established cut-off threshold vs TAPS Prescribed Medication Domain |
| between NS metric vs<br>TAP Tools | Table 6.1.2 | CP | Confusion Table for NS metric with established cut-off threshold vs TAPS Prescribed Medication Domain, by gender |
| | Figure 6.1.3 | CP | NS metric ROC curve for discriminating high risk vs low risk opioid misuse patients (defined by TAPS) |
| | Figure 6.1.4 | СР | NS metric ROC curve for discriminating high risk vs low risk opioid misuse patients (defined by TAPS), by gender |
| | Table 6.1.5 | СР | Summary of AUC of ROC curve, for NS metric vs TAPS |
| | Table 6.1.6 | CP | Summary of AUC of ROC curve, for NS metric vs TAPS by gender |
| | Table 6.1.7 | СР | Summary of Kappa Coefficient and Correlation<br>Analysis Results, NS metric vs TAP Tools |
| | Table 6.1.8 | CP | Summary of Kappa Coefficient and Correlation<br>Analysis Results, NS metric vs TAP Tools, by<br>gender |
| | Table 6.1.9 | СР | Summary of ordinal logit regression results, NS metric vs TAP Tools |
| | Table 6.1.10 | CP | Summary of ordinal logit regression results, NS metric vs TAP Tools, by gender |
| Results for<br>Exploratory Aim 2 – | Table 6.2.1 | CP | Confusion Table for NS metric with established cut-off threshold vs POMI |
| explore association between NS metric vs | Table 6.2.2 | CP | Confusion Table for NS metric with established cut-off threshold vs POMI, by gender |
| POMI Tools | Figure 6.2.3 | CP | NS metric ROC curve for discriminating high risk vs low risk opioid misuse patients (defined by POMI) |
| | Figure 6.2.4 | СР | NS metric ROC curve for discriminating high risk vs low risk opioid misuse patients (defined by POMI), by gender |
| | Table 6.2.5 | СР | Summary of AUC of ROC curve, for NS metric vs POMI |
| | Table 6.2.6 | СР | Summary of AUC of ROC curve, for NS metric vs POMI by gender |
| | Table 6.2.7 | СР | Summary of Kappa Coefficient and Correlation<br>Analysis Results, NS metric vs POMI |
| | Table 6.2.8 | СР | Summary of Kappa Coefficient and Correlation<br>Analysis Results, NS metric vs POMI, by gender |

| Section | Table/Figure | Analysis<br>Population | Title |
|---|---|---|---|
| | Table 6.2.9 | СР | Summary of ordinal logit regression results, NS metric vs POMI |
| | Table 6.2.10 | СР | Summary of ordinal logit regression results, NS metric vs POMI, by gender |
| Results for<br>Exploratory Aim 2 – | Table 6.3.1 | СР | Confusion Table for NS metric with established cut-off threshold vs OESWD |
| explore association<br>between NS metric vs | Table 6.3.2 | СР | Confusion Table for NS metric with established cut-off threshold vs OESWD, by gender |
| OESWD | Figure 6.3.3 | СР | NS metric ROC curve for discriminating high risk vs low risk opioid misuse patients (defined by OESWD) |
| | Figure 6.3.4 | СР | NS metric ROC curve for discriminating high risk vs low risk opioid misuse patients (defined by OESWD), by gender |
| | Table 6.3.5 | СР | Summary of AUC of ROC curve, for NS metric vs OESWD |
| | Table 6.3.6 | СР | Summary of AUC of ROC curve, for NS metric vs OESWD by gender |
| | Table 6.3.7 | СР | Summary of Kappa Coefficient and Correlation<br>Analysis Results, NS metric vs OESWD |
| | Table 6.3.8 | СР | Summary of Kappa Coefficient and Correlation<br>Analysis Results, NS metric vs OESWD, by<br>gender |
| | Table 6.3.9 | СР | Summary of ordinal logit regression results, NS metric vs OESWD |
| | Table 6.3.10 | СР | Summary of ordinal logit regression results, NS metric vs OESWD, by gender |
| Results for Subgroup<br>Comparison | Table 7.1 | СР | Summary table that compares selected cut-off threshold values with NS metric between 2 gender subgroups. |
| | Table 7.2 | СР | Summary table that compares discrimination ability of NS metrics with established cut-off threshold between 2 gender subgroups, with WHO ASSIST as gold standard. |
| | Table 7.3 | СР | Summary table that compares discrimination ability of TAPS tool between 2 gender subgroups, with WHO ASSIST as gold standard. |
| | Table 7.3 | СР | Summary table that compares between metrics association of NS metrics vs 1)WHO ASSIST 2) TAPS 3) OESWD 4) POMI, between 2 gender subgroups |
| <b>Protocol Deviations</b> | Table 8.1 | СР | Summary of Protocol Deviations in Study<br>Completers |
| | Listing 8.2 | CP | Listing of Protocol Deviations in Study |

| Section | Table/Figure # | Analysis<br>Population | Title |
|---------|----------------|------------------------|------------|
| | | | Completers |

## REFERENCES

- 1. Humeniuk R, Ali R. Validation of the Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) and Pilot Brief Intervention: A Technical Report of Phase II Findings of the WHO ASSIST Project. Geneva: WHO;2006.
- 2. McNeely J, Wu LT, Subramaniam G, et al. Performance of the Tobacco, Alcohol, Prescription Medication, and Other Substance Use (TAPS) Tool for Substance Use Screening in Primary Care Patients. *Annals of internal medicine*. 2016;165(10):690-699.
- 3. McNeely J, Strauss SM, Rotrosen J, Ramautar A, Gourevitch MN. Validation of an audio computer-assisted self-interview (ACASI) version of the alcohol, smoking and substance involvement screening test (ASSIST) in primary care patients. *Addiction*. 2016;111(2):233-244.
- 4. Knisely JS, Wunsch MJ, Cropsey KL, Campbell ED. Prescription Opioid Misuse Index: A brief questionnaire to assess misuse. *Journal of Substance Abuse Treatment*. 2008;35(4):380-386.
- 5. Fernandez AC, Bush C, Bonar EE, Blow FC, Walton MA, Bohnert ASB. Alcohol and Drug Overdose and the Influence of Pain Conditions in an Addiction Treatment Sample. *Journal of addiction medicine*. 2019;13(1):61-68.
- 6. Kroenke K, Spitzer RL, Williams JBW. The Patient Health Questionnaire-2: Validity of a Two-Item Depression Screener. *Medical Care*. 2003;41(11):1284-1292.
- 7. Luo X, George ML, Kakouras I, et al. Reliability, validity, and responsiveness of the short form 12-item survey (SF-12) in patients with back pain. *Spine*. 2003;28(15):1739-1745.
- 8. Keller S, Bann CM, Dodd SL, Schein J, Mendoza TR, Cleeland CS. Validity of the brief pain inventory for use in documenting the outcomes of patients with noncancer pain. *Clin J Pain*. 2014;20(5):309-319.
- 9. Cawley G, Talbot N. On Over-fitting in Model Selection and Subsequent Selection Bias in Performance Evaluation. *J Mach Learn Res.* 2010;11:2079-2107.
- 10. Youngstrom EA. A Primer on Receiver Operating Characteristic Analysis and Diagnostic Efficiency Statistics for Pediatric Psychology: We Are Ready to ROC. *Journal of Pediatric Psychology*. 2014;39(2):204-221.
- 11. Cohen J. A Coefficient of Agreement for Nominal Scales. *Educational and Psychological Measurement.* 1960;20(1):37-46.
- 12. Landis JR, Koch GG. The measurement of observer agreement for categorical data. *Biometrics*. 1977;33(1):159-174.
- 13. Kendall MG. Rank correlation methods London: Griffin; 1970.
- 14. McCullagh P. Regression Models for Ordinal Data. *Journal of the Royal Statistical Society: Series B (Methodological)*. 1980;42(2):109-127.
- 15. Rubin D. *Multiple imputation for nonresponse in surveys* Vol 81. Hoboken, NJ: John Wiley & Sons; 2004.